CLINICAL TRIAL: NCT00579566
Title: Novel Biochemical and Molecular Determinants for Soft Tissue Sarcoma
Status: Recruiting | Type: Observational
Sponsor: Memorial Sloan Kettering Cancer Center (Other)
Responsible Party: Sponsor
Other Study IDs: 02-060
Record Dates: First submitted 2007-12-19; First posted 2007-12-24 (Estimated); Last update posted 2025-07-30 (Actual); Status verified 2025-07

CONDITIONS: Sarcoma
Keywords: Biochemical Determinants; Molecular Determinants
MeSH Terms: conditions — Sarcoma

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Tissue, Blood
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- 1: Sarcoma patients undergoing core biopsy, incisional biopsy or definitive surgical resection for soft tissue masses of extremity, trunk or retroperitoneum
  Interventions: Other: Specimen protocol

INTERVENTIONS:
Other: Specimen protocol — The research specimen will be obtained from the residual specimen that would otherwise be discarded per usual hospital procedure.

SUMMARY:
The purpose of this study is to study normal and sarcoma cells. To study these cells we need to have human tissue. You will be having or have already had a procedure to remove tissue. We would like to use some of this tissue. We will use it for laboratory studies on the diagnosis,behavior and treatment of sarcoma. We will perform an extensive analysis of your samples. We will only use extra tissue left over after all needed testing has been done or remove an additional small amount of tissue if you are having a biopsy. We will also take blood samples before and/or after your procedure to measure biochemical factors that may help us predict the behavior of sarcoma.

DETAILED DESCRIPTION:
In this protocol, we plan to identify specific markers from biochemical, proteomic, epigenetic and molecular genetic analyses that predict clinical outcome, responsiveness to therapy and might serve as promising therapeutic targets in patients with soft tissue sarcoma.

ELIGIBILITY:
Inclusion Criteria:

* All patients with known or suspected sarcoma who will have or have had tissue removed for therapeutic or diagnostic purposes.
* Patients will be entered without preference for any particular racial/ethnic group or gender.
* Patients may have received prior hormonal therapy, cytotoxic chemotherapy, irradiation, immunotherapy or surgical therapy.
* Tissue specimens must be large enough in quantity to allow routine pathologic analysis, with the research laboratory specimen removed from the residual specimen, which would otherwise be discarded. Optimal tissue amounts for snap freeze: Core biopsy - 2 tissue cores Incisional biopsy- 0.5 to 1.5 grams Resected sarcoma specimen- 1.0 to 50 grams depending on size of specimen Normal fat or muscle tissue - 0.5 to 4.0 grams (if available from resected sarcoma specimen) Optimal tissue amounts for RNA later Core biopsy - 2 tissue cores Incisional biopsy- 30 mg (three 3 x 3 x 3 mm cubes) Resected sarcoma specimen - 30 mg (three 3 x 3 x 3 mm cubes) Normal fat or muscle tissue - 30 mg (three 3 x 3 x 3 mm cube

Exclusion Criteria:

- None

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients seen or referred by Memorial Sloan-Kettering Cancer physicians
Sampling Method: Non-Probability Sample
Enrollment: 3000 (Estimated)
Dates: Start 2002-06 (Actual); Primary Completion 2026-06 (Estimated); Study Completion 2026-06 (Estimated)

PRIMARY OUTCOMES:
establish and maintain a specimen bank and sarcoma cell line resource | 2 years
  for laboratory-based studies on the causes, prevention, diagnosis and treatment of human soft tissue sarcoma

SECONDARY OUTCOMES:
identify new rational therapeutic targets | 2 years

CONTACTS AND LOCATIONS:
Overall Officials: Singer Singer, MD, Principal Investigator — Memorial Sloan Kettering Cancer Center
Locations (7):
- United States (7):
  - Memorial Sloan Kettering Basking Ridge (Consent and Follow-Up), Basking Ridge, New Jersey
  - Memorial Sloan Kettering Monmouth (Consent and Followup), Middletown, New Jersey
  - Memorial Sloan Kettering Bergen (Consent and Follow up), Montvale, New Jersey
  - Memorial Sloan Kettering Commack (Consent and Follow-Up), Commack, New York
  - Memorial Sloan Kettering Westchester (Consent and Followup), Harrison, New York
  - Memorial Sloan Kettering Cancer Center (All Protocol Activities), New York, New York
  - Memorial Sloan Kettering Nassau (Consent and Followup), Rockville Centre, New York

REFERENCES:
- See also: Memorial Sloan Kettering Cancer Center — http://www.mskcc.org